CLINICAL TRIAL: NCT05295121
Title: An Open-label, Randomized, Cross-over Study With 2 Treatments (Fasting and After Meals), 3 Periods, 2 Sequences, and an Adaptive, Two-stage Design to Evaluate the Effect of Food Intake on the Bioavailability of XC221 100 mg Tablets at a Single Dose in Healthy Volunteers
Brief Title: Study of the Effect of Food Intake on the Bioavailability of XC221 100 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XC221-01-04-2021
Record Dates: First submitted 2022-01-28; First posted 2022-03-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — XC221

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC221, fasted (Experimental): Administration of XC221 in fasted state in Dosing Periods 1 and 2 followed by administration of XC221 in fasted state in Dosing Period 3
  Interventions: Drug: XC221 100 mg tablets
- XC221, fed (Experimental): Administration of XC221 in fed state in Dosing Periods 1 and 2 followed by administration of XC221 in fasted state in Dosing Period 3
  Interventions: Drug: XC221 100 mg tablets

INTERVENTIONS:
Drug: XC221 100 mg tablets — XC221, 3 discrete doses separated by 7-day wash-out periods

SUMMARY:
Primary objective of the study: evaluation of the effect of food intake on the bioavailability of XC221 100 mg tablets after a single oral administration in fed or fasted condition.

Additional objective of the study: evaluation of pharmacokinetic parameters, safety and tolerability of XC221 100 mg tablets in healthy volunteers after single oral administration in fed or fasted condition.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers aged 18 to 45 years (inclusive).
2. Presence of written consent of the volunteer to participate in the study in accordance with applicable law.
3. Body mass index (BMI) within the range of 18.5 ≤ BMI ≤ 30 kg/m2 with a body weight not less than 45 kg and not more than 100 kg.
4. Verified diagnosis "healthy": no deviations from the reference values of the data of standard clinical, laboratory and instrumental methods of examination.
5. The consent of the volunteer (including the partner) to use adequate methods of contraception during the study and 3 weeks after its completion.
6. Hemodynamic and other vital signs within normal limits (reference intervals are 60-90 bpm at rest for heart rate (HR), 16-20 breaths/min for respiratory rate (RR), 35.5 to 36.9°C for body temperature, normal blood pressure (BP) is considered to be systolic blood pressure (SBP) in the range of 110-130 mmHg; diastolic blood pressure (DBP) is 60-85 mmHg).

Exclusion Criteria:

1. Hypersensitivity to the active substance XC221 (N-[2-(1H-imidazol-4-yl)-ethyl]-6-oxo-δ-lactam) and/or any other component of the drug product.
2. A history of allergy.
3. A history of bronchial asthma, recurrent nasal or paranasal sinus polyposis, allergic rhinitis.
4. Hereditary lactose intolerance, lactase deficiency and glucose-galactose malabsorption syndrome.
5. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine, digestive, urinary, hematopoietic, immune and musculoskeletal systems, mental illness in the history.
6. Acute infectious diseases (including influenza, acute respiratory infections) within 30 days prior to the study.
7. Surgical interventions on the gastrointestinal tract in the anamnesis (except appendectomy).
8. Taking any medications, including vitamins, herbal preparations, and dietary supplements within 14 days prior to screening.
9. Taking medications that have significant effects on hemodynamics or liver function (barbiturates, omeprazole, cimetidine, etc.) for less than 30 days before screening.
10. Vital signs outside the reference intervals: SBP less than 110 mmHg or greater than 130 mmHg; DBP less than 60 mmHg or greater than 85 mmHg; HR less than 60 bpm or greater than 90 bpm; body temperature less than 35.5 or greater than 36.9° C, RR less than 16 or greater than 20 bpm.
11. Laboratory values outside the reference intervals.
12. Intake of more than 10 units of alcohol per week (where each unit equals 30 ml of spirits or 120 ml of wine or 330 ml of beer) or anamnestic evidence of alcoholism, drug addiction, substance abuse, drug abuse.
13. Smoking more than 10 cigarettes per day and failure to abstain from smoking 48 hours before the study and during the hospital stay.
14. Special diet (e.g., vegetarian, vegan, restricted salt intake) or lifestyle (night work, extreme physical activity).
15. Consumption of alcohol, caffeine, and xanthine-containing products 72 hours before taking the drug product.
16. Consumption of citrus fruits, cranberries and products containing them, preparations or products containing St. John's wort - 7 days before taking the IP. 17.
17. Dehydration due to diarrhea, vomiting, or other reason within the last 24 hours prior to IP administration.
18. Positive result of examination for antibodies to HIV type 1 and 2, syphilis, markers of hepatitis B and C.
19. Positive result of rapid test for COVID-19.
20. Positive breath alcohol test.
21. Positive urine drug test (cocaine, marijuana, amphetamine, methamphetamine, morphine, barbiturates).
22. Pregnancy, breastfeeding, positive urine pregnancy test (for women of preserved reproductive potential).
23. Use of hormonal contraceptives (oral, transdermal, injectable, implantable) by a female volunteer for 2 months prior to the drug administration.
24. Donation of blood (450 ml or more) within 30 days prior to the study.
25. Participation in a clinical drug study of any phase within 90 days prior to the start of the study.
26. Unavailability for observation during the study, inability to keep the visit schedule, inability to be hospitalized for the required duration, high likelihood of problems with successful insertion of a venous catheter or performing a forearm vein puncture.
27. Belonging to a vulnerable group of volunteers (minors; incapacitated; people with limited free will or possibly participating under compulsion (serving a sentence in prison, being in custody in detention centers, military personnel)), as well as law enforcement officers.
28. Other reasons that, in the opinion of the researcher, prevent the participation of the volunteer in the research or create an unreasonable risk.

Withdrawal criteria:

1. Withdrawal of consent to participate in the study.
2. SAE, irrespective of causal relationship to drug intake.
3. Any other AE if the researcher believes it is in the best interest of the volunteer to discontinue participation in the study.
4. Missing two consecutive or four or more blood sampling points to determine pharmacokinetic parameters during the same period of the pharmacokinetics study.
5. Violation of study protocol requirements (including because the volunteer refuses to cooperate with the investigator, is late to the clinic, etc.).
6. Volunteer is undergoing or requires treatment that may affect the pharmacokinetic parameters of the drug.
7. Volunteer requires inpatient treatment while participating in the study.
8. Vomiting and/or diarrhea in volunteer within 24 hours prior to the drug administration or within 3 hours (2 maximum Tmax for XC221) after the drug administration.
9. Positive urine drug test result.
10. Positive breath alcohol test.
11. Positive urine pregnancy test.
12. Positive test for COVID-19.
13. Discontinuation of the study at the discretion of the Sponsor or regulatory agency.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 12 hours after dosing on Day 1, Day 8, and Day 15
  Maximum plasma concentration (Cmax) of XC221GI (active ingridient) and XC221A (metabolite)
Pharmacokinetics - AUC0-t | From 0 to 12 hours after dosing on Day 1, Day 8, and Day 15
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t) of XC221GI (active ingridient) and XC221A (metabolite)
Pharmacokinetics - AUC0-inf | From 0 to 12 hours after dosing on Day 1, Day 8, and Day 15
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) of XC221GI (active ingridient) and XC221A (metabolite)

SECONDARY OUTCOMES:
Safety and Tolerability: adverse event (AE) number and frequency | From the screening (and signing informed consent form) to Day 16 of the study or to an early termination visit within the time frame of the study (from Day -1 to Day 16)
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: adverse event (AE) characteristics | From the screening (and signing informed consent form) to Day 16 of the study or to an early termination visit within the time frame of the study (from Day -1 to Day 16)
  Description and severity of AEs or serious AEs (SAEs), concomitant therapy for AEs/SAEs, causal relationship with XC221, outcomes.
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, from Day -1 to Day 2, from Day 7 to Day 9, from Day 14 to Day 16 and/or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, from Day -1 to Day 2, from Day 7 to Day 9, from Day 14 to Day 16 and/or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, from Day -1 to Day 2, from Day 7 to Day 9, from Day 14 to Day 16 and/or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, from Day -1 to Day 2, from Day 7 to Day 9, from Day 14 to Day 16 and/or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, from Day -1 to Day 2, from Day 7 to Day 9, from Day 14 to Day 16 and/or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, from Day -1 to Day 2, from Day 7 to Day 9, from Day 14 to Day 16 and/or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Physical examination results
Safety and Tolerability: urinalysis - color | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  pH of the urine
Safety and Tolerability: urinalysis - specific gravity | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Specific gravity of the urine
Safety and Tolerability: urinalysis - nitrites | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Nitrites in the urine (+/-)
Safety and Tolerability: urinalysis - protein | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - glucose | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis - ketones | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Ketones in the urine (mmol/L)
Safety and Tolerability: urinalysis - urobilinogen | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Urobilinogen in the urine (mmol/L)
Safety and Tolerability: urinalysis - bilirubin | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Bilirubin in the urine (+/-)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  White blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - cylinders (except hyaline) | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Cylinders (except hyaline) in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - bacteria | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Bacteria in the urine (number in sight)
Safety and Tolerability: complete bood count - hemoglobin | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Hemoglobin, g/dL
Safety and Tolerability: complete bood count - red blood cells | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Red blood cells, 10^6/uL
Safety and Tolerability: complete bood count - hematocrit | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Hematocrit, %
Safety and Tolerability: complete bood count - platelets | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Platelets, 10^3/uL
Safety and Tolerability: complete bood count - white blood cells | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  White blood cells, 10^3/uL
Safety and Tolerability: complete bood count - erythrocyte sedimentation rate | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete bood count - neutrophils | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Neutrophils, %
Safety and Tolerability: complete bood count - lymphocytes | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Lymphocytes, %
Safety and Tolerability: complete bood count - eosinophils | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Eosinophils, %
Safety and Tolerability: complete bood count - monocytes | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Monocytes, %
Safety and Tolerability: complete bood count - basophils | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Basophils, %
Safety and Tolerability: blood test results - total protein | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - creatinine | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - urea | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Urea in blood serum, mmol/L
Safety and Tolerability: blood test results - glucose | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total bilirubin | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - direct bilirubin | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Direct bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - total cholesterol | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - triglycerides | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  Triglycerides in blood serum, mmol/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  AST in blood serum, U/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  ALP in blood serum, U/L
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | Screening and Day 16 or on early termination visit within the time frame of the study (from Day -1 to Day 16)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company "Research Center Eco-Safety", Saint Petersburg, Russia